CLINICAL TRIAL: NCT02636179
Title: Evaluation of the Prevalence of Asthma in a Cohort of Children Born After In Vitro Fertilization (Aged 11-15) Compared With Spontaneously Conceived Children of the Same Age Range
Brief Title: Evaluation of the Prevalence of Asthma in a Cohort of Children Born After IVF (Aged 11-15) Compared With a Control Group
Acronym: EMCeFIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Principal Investigator, Pierre Boyer, Head of Assisted Reproductive Technologies Laboratory, Hospital St. Joseph, Marseille, France
Other Study IDs: RCB 2015-A00997-42
Record Dates: First submitted 2015-12-14; First posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Asthma
Keywords: In Vitro Fertilization, follow-up of children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 448 children: Children aged 11-15 years from a historical cohort born after In Vitro Fertilization or Intracytoplasmic Sperm Injection at Hospital Saint Joseph of Marseille
  Interventions: Other: Comparative epidemiological survey
- 1344 children: Children aged 11-15 years born spontaneously schooling in the same geographic area as case
  Interventions: Other: Comparative epidemiological survey

INTERVENTIONS:
Other: Comparative epidemiological survey — The method used to select the control group will be the random sampling of eligible schools. It will be defined according to the place of schooling of the historic cohort of children. The children will be matched as close as possible based on sex, age, school class and type of school (public/private).

SUMMARY:
Assisted Reproduction Technologies (ART) are increasingly being used worldwide as a result of fertility decline likely caused by changes in both environment and social behaviour. Considering this large usage, it is important to evaluate the potential risk on the health of children conceived using ART.

According to the literature, children born after ART are more likely to be at higher risk of health problems than spontaneously conceived ones. Interestingly, recent studies suggested an increase of asthma prevalence in children conceived using In Vitro Fertilization (IVF).

The purpose of this study is to evaluate the prevalence of asthma in school adolescents from a cohort of children born after In Vitro Fertilization (IVF), aged 11-15 years as compared to a control group composed of the same age range spontaneously conceived individuals.

The expected outcome of this study will provide new information regarding these children to ART professionals of and to their own families, by focusing on an age range (between 11 and 15 years) for which very little information is available to date.

DETAILED DESCRIPTION:
The methodology is a comparative epidemiological survey, between children from a historical cohort born after intraconjugal In Vitro Fertilization (singleton or twin) aged 11-15 years and a control group recruited in schools after the agreement of Academic Inspection.

Parents of the two groups will be contacted either by phone calls or through written information given in the schools. They will receive the questionnaire and an information letter, once they give their agreement to be a part of the study.

Data collection will be conducted using two anonymous questionnaires. The first questionnaire was built based on items proposed in the international Health Behaviour in School-aged Children (HBSC) survey of the World Health Organization (WHO). The second questionnaire will be sent to parents. It will focus on the pregnancy and it will be used to adjust the analysis.

This study was submitted and approved by an Institutional Review Board in France (Comité de Protection des Personnes Sud-Méditerranée II) on 11th September 2015.

ELIGIBILITY:
Inclusion Criteria:

* Case :
* Children conceived by Intraconjugal In Vitro Fertilization/Intracytoplasmic Sperm Injection treatment
* Children aged 11-15 years
* Singleton and twins
* School children
* Control :
* Children born spontaneously (without IVF)
* Children aged 11-15 years
* Children in the same place of schooling of the case

Exclusion Criteria:

* Case :
* Children not born by Intraconjugal In Vitro Fertilization/Intracytoplasmic Sperm Injection treatment (donor)
* Children whose parents refuse the participation
* Triplet and more pregnancies
* Children who cannot attend ordinary school
* Children from families where an infant has passed away
* When the participation agreement was not signed
* Control :
* Children whose parents have benefited ART
* When the participation agreement was not signed
* Children whose aged and sex are unknown
* Triplet and more pregnancies

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The investigators will include children born after In Vitro Fertilization/Intracytoplasmic Sperm Injection treatment from a historic cohort and children born spontaneously (without ART), attending schools in the same geographic area as IVF/ICSI children. Parents will be contacted before to include children.
Sampling Method: Non-Probability Sample
Enrollment: 1792 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-01 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of asthma | 15 month
  (will be assessed using the questionnaire of international Health Behaviour in School-aged Children [HBSC] survey).

SECONDARY OUTCOMES:
Prevalence of chronic diseases other than asthma | 15 month
  (will be assessed using the questionnaire of international Health Behaviour in School-aged Children [HBSC] survey)
Physical well-being | 15 month
  (will be assessed using the questionnaire of international Health Behaviour in School-aged Children [HBSC] survey)
Anthropometric measures | 15 month
  (will be assessed using the questionnaire of international Health Behaviour in School-aged Children [HBSC] survey)
Age of puberty in girls | 15 month
  (will be assessed using the questionnaire of international Health Behaviour in School-aged Children [HBSC] survey)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint Joseph de Marseille, Marseille, France

REFERENCES:
- [Background] Anzola AB, Pauly V, Geoffroy-Siraudin C, Gervoise-Boyer MJ, Montjean D, Boyer P. The first 50 live births after autologous oocyte vitrification in France. J Assist Reprod Genet. 2015 Dec;32(12):1781-7. doi: 10.1007/s10815-015-0603-2. Epub 2015 Oct 30. PMID 26519416
- [Background] Meddeb L, Boyer M, Pauly V, Tourame P, Rossin B, Pfister B, Boyer P. [Procedure used to follow-up a cohort of IVF children. Interests and limits of tools performed to longitudinal follow up for a monocentric cohort]. Rev Epidemiol Sante Publique. 2011 Apr;59(2):97-105. doi: 10.1016/j.respe.2010.11.004. Epub 2011 Mar 22. French. PMID 21429679